CLINICAL TRIAL: NCT06937112
Title: Clinical Application of a Novel 18F Labeled Fibroblast Activation Protein (FAP) Targeted Molecular Probe in Early Tumor Diagnosis
Brief Title: 18F Labeled FAP Targeted Molecular Probe in Early Tumor Diagnosis
Status: Recruiting | Type: Observational
Sponsor: Nanjing First Hospital, Nanjing Medical University (Other)
Responsible Party: Principal Investigator, Feng Wang, Chief physician, Nanjing First Hospital, Nanjing Medical University
Other Study IDs: KY20250407-KS-1
Record Dates: First submitted 2025-04-18; First posted 2025-04-22 (Actual); Last update posted 2025-04-22 (Actual); Status verified 2025-04

CONDITIONS: Lung Cancers; Pancreatic Cancer; Neuroendocrine Tumors; Thyroid Cancer
MeSH Terms: conditions — Lung Neoplasms; Pancreatic Neoplasms; Neuroendocrine Tumors; Thyroid Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PET-CT examination — Intravenous injection of 18F-FAPI-YQ104 for PET-CT examination

SUMMARY:
Evaluate the safety of the novel FAP targeted molecular probe 18F-FAPI-YQ104 labeled with radioactive isotopes in clinical applications and verify its effectiveness in tumor diagnosis.

ELIGIBILITY:
Inclusion Criteria:

- 1. Volunteer for the trial, with the patient or their legal guardian signing the informed consent form; 2. Volunteers are not limited by gender, and the age range is from 18 to 75 years old, including both ends; 3. Other imaging examination methods (CT, MRI, etc.) revealed tumor occupying lesions; 4. Patients with lung cancer, thyroid cancer, pancreatic cancer, melanoma, and neuroendocrine tumors who can obtain the final pathological results.

5. Kidney: GFR > 50 ml/min, ERPF > 280 ml/min, platelet count (PLT) > 75,000/μL, white blood cell (WBC) > 3,000/μL, alanine aminotransferase (ALT) and aspartate aminotransferase (AST) levels less than 3 times the normal value.

Exclusion Criteria:

* 1. Individuals with a history of allergies to similar drugs (drugs with similar chemical or biological components to FAPI), allergic constitution, or current allergic diseases; 2. Those who are currently conducting clinical research on other drugs or have participated in any clinical research on drugs (excluding vitamins and minerals); 3. There are other clinical problems that are difficult to control (such as HIV, hepatitis C virus infection or active hepatitis B, or other serious chronic infections and serious mental, neurological, cardiovascular, respiratory and other system diseases); 4. Red blood cell RBC<4 × 1012, white blood cell WBC<3 × 109, hemoglobin<110g/L, PLT<75000×109； 5. Significant abnormalities in liver and kidney function, with GFR less than 50 ml/min; 6. Tumor burden greater than 50%, or significant spinal cord compression; 7. Expected survival period is less than six months; Chemotherapy within June; 8. Having severe acute comorbidities or severe refractory mental disorders; 9. Pregnant and lactating women (where pregnancy is defined as a positive urine pregnancy study); 10. Patients whose physical condition is not suitable for radiation examination; 11. Other situations that researchers consider unsuitable for participating in the experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants were recruited through hospital electronic records and community health centers
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
SUVmax of lesion uptake value | 60 minutes after administration

CONTACTS AND LOCATIONS:
Locations (1):
- Nanjing First Hospital, Nanjing, Jiangsu, China